CLINICAL TRIAL: NCT00806468
Title: A Double Blind, Placebo Controlled, Randomized, Monocentre Cross-over Study to Investigate the Effect of Desmopressin on the Nocturnal Micturition Frequency in Patients With Parkinson Disease
Brief Title: Effect of Desmopressin on the Nocturnal Micturition Frequency in Patients With Parkinson Disease
Acronym: DEPOPA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: PD Dr. Thomas Vogt, Johannes Gutenberg University Mainz, Department of Neurology
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DEPOPA-2008
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2010-12-20 (Estimated); Status verified 2010-06

CONDITIONS: Parkinson Disease
Keywords: nycturia; Parkinson syndrome; desmopressin; Nocturnal polyuria in patients with Parkinson syndrome
MeSH Terms: conditions — Parkinson Disease; Nocturia | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Desmopressin (Experimental): Desmopressin 0,2 mg once daily and Desmopressin 0,2 mg bid for one week each.
  Interventions: Drug: Desmotabs

INTERVENTIONS:
Drug: Desmotabs — Desmotabs encapsulated, 0,2 mg once daily for one week, 0,2 mg bid for one week

SUMMARY:
This study will be conducted to study the effect of Desmopressin on the nocturnal micturition frequency in patients with idiopathic Parkinson syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with idiopathic Parkinson Syndrome
* 18 to 85 years
* Nocturnal Pollakisuria > 2 mictions /night (documented in Screening phase )
* Na+ i.S > 135 mmol/l
* Patient is able to understand all aspects and individual consequences of the clinical trial
* An informed consent signed and dated by the patient is available prior to any study specific treatment
* The study is consistent with the patients´ request for an appropriate treatment

Exclusion Criteria:

* Intake of the following concomitant medication: Carbamazepin, Oxcarbazepine, diuretics (Furosemide, Torasemide), non steroidal antiphlogistics, Loperamide, antidiuretic hormone analoga (besides study medication), drugs for treatment of bladder disfunction, in particular anticholinergics
* Central Diabetes insipidus
* Known heart insufficiency (NYHA Stad. III und IV)
* clinical relevant kidney insufficiency
* Habitual and psychogenic Polydipsia
* Hypersensitivity or allergy against the trial medication or any other ingredient of the trial medication
* Participation in another clinical trial during or within 6 months prior to this clinical trial
* Medical or psychological condition, which might endanger the proper conduction of the clinical trial
* Known drug or alcohol abuse

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-02; Primary Completion 2010-12 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
average nocturnal micturition frequency within the 2 weeks treatment phase each | 6 weeks

SECONDARY OUTCOMES:
safety and efficacy on nocturnal micturition frequency of Desmopressin in patients with Parkinson syndrome | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Vogt, MD, Principal Investigator — Johannes Gutenberg University Mainz, Department of Neurology
Locations (1):
- Klinikum der Johannes Gutenberg-Universität Mainz, Studienzentrum Neurologie, Langenbeckstr. 1, 55131 Mainz, Mainz, Germany